CLINICAL TRIAL: NCT01715857
Title: A Multicenter Registry on the Clinical Practice of Inhalation Anesthesia With Sevoflurane in China
Brief Title: Clinical Practice of Inhalation Anesthesia With Sevoflurane in China
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P13-934
Record Dates: First submitted 2012-09-02; First posted 2012-10-29 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Anesthesia, General
Keywords: Economics, Pharmaceutical; Physician's Practice Patterns; Chinese; Sevoflurane

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chinese Patients Requiring Surgery with Sevoflurane Anesthesia: Participants who were scheduled for surgery requiring sevoflurane anesthesia with endotracheal intubation or laryngeal mask airway (LMA) per approved product information of sevoflurane in China

SUMMARY:
Until recently, there was a lack of understanding and consensus among Chinese anesthesiologists how they should practice general anesthesia with volatile anesthetics, since there was no standard of inhalation practice. In August 2011, the Anesthesiology branch of the Chinese Medical Association launched the first version of Chinese Consensus of Standard Clinical Practice for Inhalation Anesthesia (Consensus) in order to standardize the practice in China.

The proposed registry is aimed to evaluate the current inhalation practice one year after the Consensus has been released, and related patient outcome. This registry evaluated sevoflurane anesthesia, including screening, induction, maintenance, emergence, and follow-up within 24 hours post-operation.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman, aged from 18 to 70 years old.
2. American Society of Anesthesiologists (ASA) physical status: I, II and III.
3. Surgery requiring sevoflurane anesthesia with endotracheal intubation or laryngeal mask airway (LMA).
4. The type of surgery is either general surgery, or orthopedics, or gynecology.
5. The duration of anesthesia ranges from 1 to 5 hours.

Exclusion Criteria:

1. History of clinically significant cardiovascular, pulmonary, renal, hepatic or central nervous system or muscle disease.
2. Known hypersensitivity or history of unusual response to any halogenated anesthetics.
3. Personal or familial history of malignant hyperthermia.
4. Female patients who are either pregnant or breast feeding.
5. General anesthesia is administered with total intravenous anesthesia (TIVA) of propofol or sevoflurane maintenance combined with propofol continuous infusion during maintenance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients undergoing surgery require general anesthesia (sevoflurane) with endotracheal intubation or laryngeal mask.
Sampling Method: Non-Probability Sample
Enrollment: 4100 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yue Kang, MD, Study Director — AbbVie
Locations (36):
- China (36):
  - Site Reference ID/Investigator# 84317, Beijing
  - Site Reference ID/Investigator# 86755, Beijing
  - Site Reference ID/Investigator# 96155, Beijing
  - Site Reference ID/Investigator# 84320, Beijing
  - Site Reference ID/Investigator# 84316, Beijing, Xicheng District
  - Site Reference ID/Investigator# 84321, Changchun, Jilin
  - Site Reference ID/Investigator# 86754, Changchun, Jilin
  - Site Reference ID/Investigator# 86764, Changsha, Hunan
  - Site Reference ID/Investigator# 86767, Changsha, Hunan
  - Site Reference ID/Investigator# 100206, Chengdu
  - Site Reference ID/Investigator# 86762, Chongqing
  - Site Reference ID/Investigator# 84338, Guangzhou
  - Site Reference ID/Investigator# 106416, Guangzhou
  - Site Reference ID/Investigator# 84337, Guangzhou
  - Site Reference ID/Investigator# 102457, Guangzhou
  - Site Reference ID/Investigator# 84333, Guangzhou, Guangdong
  - Site Reference ID/Investigator# 100095, Guangzhou, Guangdong
  - Site Reference ID/Investigator# 84334, Harbin, Heilongjiang
  - Site Reference ID/Investigator# 86759, Jinan, Shandong
  - Site Reference ID/Investigator# 84318, Kunming, Yunnan
  - Site Reference ID/Investigator# 86757, Kunming, Yunnan
  - Site Reference ID/Investigator# 84336, Lanzhou, Gansu
  - Site Reference ID/Investigator# 84322, Lanzhou, Gansu
  - Site Reference ID/Investigator# 86761, Nanchang, Jiangxi
  - Site Reference ID/Investigator# 102455, Qingdao
  - Site Reference ID/Investigator# 78434, Shanghai
  - Site Reference ID/Investigator# 86073, Shanghai
  - Site Reference ID/Investigator# 84342, Shanghai
  - Site Reference ID/Investigator# 84314, Shenyang, Liao Ning
  - Site Reference ID/Investigator# 84319, Shijiazhuang Hebei
  - Site Reference ID/Investigator# 100207, Tianjin
  - Site Reference ID/Investigator# 95295, Tianjin
  - Site Reference ID/Investigator# 86760, Wuhan, Hubei
  - Site Reference ID/Investigator# 86766, Zhengzhou, Henan
  - Site Reference ID/Investigator# 86763, Zhengzhou, Henan
  - Site Reference ID/Investigator# 86769, Zunyi, Guizhou

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chinese Patients Requiring Surgery With Sevoflurane Anesthesia
Started | 4100
Completed | 4004
Not Completed | 96
Not completed — Did Not Meet Eligibility Criteria | 96

BASELINE CHARACTERISTICS:
Arm/Group | Chinese Patients Requiring Surgery With Sevoflurane Anesthesia
Number analyzed (Participants) | 4004
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.54 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2720
  Male | 1284
American Society of Anesthesiologist (ASA) Physical Status [Number; unit: percentage of participants] — ASA Physical Status Classification System: ASA Physical Status I = A normal healthy patient; ASA Physical Status II = A patient with mild systemic disease; ASA Physical Status III = A patient with severe systemic disease; ASA Physical Status IV = A patient with severe systemic disease that is a constant threat to life; ASA Physical Status V = A moribund patient who is not expected to survive without the operation; ASA Physical Status VI = A declared brain-dead patient whose organs are being removed for donor purposes
  percentage of participants
    ASA Physical Status I | 47.33
    ASA Physical Status II | 49.18
    ASA Physical Status III | 3.50
    ASA Physical Status IV | 0
    ASA Physical Status V | 0
Type of Surgery [Number; unit: percentage of participants]
  General Surgery | 55.09
  Gynecologic Surgery | 28.17
  Orthopedic Surgery | 16.73
Body Weight [Mean (Standard Deviation); unit: kilograms] | 62.19 (10.96)

OUTCOME MEASURES:

1. Primary Outcome: Anesthesiologist Satisfaction With the Anesthesia Using a Numeric Analog Scale (NAS)
Description: Anesthesiologist satisfaction with the anesthesia was recorded by the anesthesiologist at the end of the operation using a NAS from 0 (not satisfied at all) to 10 (completely satisfied). The satisfaction of induction, maintenance, and emergence accounts for 20%, 50%, and 30% of the score, respectively.
Time Frame: End of surgery
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Chinese Patients Requiring Surgery With Sevoflurane Anesthesia
Number analyzed (Participants) | 4004
scores on a scale | 9.14 (0.85)

2. Primary Outcome: Participant Satisfaction With the Anesthesia Using a Numeric Analog Scale (NAS)
Description: Participant satisfaction with the anesthesia recorded approximately 24 hours after the end of the operation using a NAS from 0 (not satisfied at all) to 10 (completely satisfied).
Time Frame: 24 hours after end of surgery
Population: All participants who received study drug and with available data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Chinese Patients Requiring Surgery With Sevoflurane Anesthesia
Number analyzed (Participants) | 4004
scores on a scale | 9.21 (0.91)

3. Secondary Outcome: Time to Eye Opening
Description: After cessation of anesthesia, the investigators lightly tapped on the participant's forehead or shoulder and asked the participant to open their eyes. This process was repeated approximately every minute until eye opening occurred.
Time Frame: From cessation of sevoflurane administration until the participant opened their eyes, up to 80 minutes
Population: All participants who received study drug and with available data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chinese Patients Requiring Surgery With Sevoflurane Anesthesia
Number analyzed (Participants) | 3982
minutes | 17.30 (11.56)

4. Secondary Outcome: Time to Extubation
Description: Time to extubation was measured from the time sevoflurane administration had stopped until tracheal extubation or laryngeal mask airway (LMA) removal occurred.
Time Frame: From cessation of sevoflurane administration until tracheal extubation occurred, up to 80 minutes
Population: All participants who received study drug and with available data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chinese Patients Requiring Surgery With Sevoflurane Anesthesia
Number analyzed (Participants) | 3981
minutes | 20.28 (13.50)

5. Secondary Outcome: Cost of Anesthetics Including Sevoflurane (Yuan Renminbi [RMB]/Hour)
Description: Cost of anesthetics is the sum of the cost of sevoflurane and other anesthetics including narcotics and muscle relaxants. Cost of sevoflurane = unit price of sevoflurane multiplied by the used volume of sevoflurane. Cost of other anesthetics = unit price of anesthetics multiplied by the total volume of anesthetics in the ampoule.
Time Frame: Anesthetic duration between 1 to 5 hours
Population: All participants who received study drug and with available data.
Measure: Mean (Standard Deviation); unit: Yuan renminbi [RMB]/hour
Arm/Group | Chinese Patients Requiring Surgery With Sevoflurane Anesthesia
Number analyzed (Participants) | 3874
Yuan renminbi [RMB]/hour | 249.79 (168.01)

6. Secondary Outcome: Non-compliance of Sevoflurane End Tidal Concentration Following the Consensus
Description: Non-compliance of sevoflurane end tidal concentration was defined as the percentage of time points for the maintenance period (excluding washout phase) that were below the sevoflurane end tidal concentration boundary of 0.6 minimal alveolar concentration (MAC) based on the Consensus. A higher percentage indicates a higher degree of non-compliance.
Time Frame: During maintenance (up to 5 hours)
Population: All participants who received study drug and with available data.
Measure: Number; unit: percentage of timepoints
Units Other Than Participants: Timepoints for Maintenance Period
Arm/Group | Chinese Patients Requiring Surgery With Sevoflurane Anesthesia
Number analyzed (Participants) | 3941
Number analyzed (Timepoints for Maintenance Period) | 44374
percentage of timepoints | 17.82

7. Secondary Outcome: Non-compliance of Sevoflurane Vaporizer Setting Following the Consensus
Description: Non-compliance of sevoflurane vaporizer setting was defined as the percentage of time points for the maintenance period outside the range of 1.0 - 1.5 minimal alveolar concentration (MAC) during the maintenance period (excluding washout phase) based on the Consensus. A higher percentage indicates a higher degree of non-compliance.
Time Frame: During maintenance (up to 5 hours)
Population: All participants who received study drug and with available data.
Measure: Number; unit: percentage of timepoints
Units Other Than Participants: Timepoints During Maintenance
Arm/Group | Chinese Patients Requiring Surgery With Sevoflurane Anesthesia
Number analyzed (Participants) | 3972
Number analyzed (Timepoints During Maintenance) | 54454
percentage of timepoints | 42.31

ADVERSE EVENTS:
Time Frame: All serious adverse events (SAEs) were required to be collected in the registry from the time the physician obtained the participant's informed consent until 30 days following treatment (approximately 31 days).
Description: Spontaneous adverse events (AEs) were also to be collected from the time the physician obtained the participant's informed consent until 30 days following treatment (total of approximately 31 days); there were no spontaneously reported AEs from the registry.
Arm/Group | Chinese Patients Requiring Surgery With Sevoflurane Anesthesia
Serious Adverse Events (participants affected / at risk) | 0/4004
Other Adverse Events (participants affected / at risk) | 0/4004

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.